CLINICAL TRIAL: NCT03535272
Title: Bismuth Subsalicylate's Role in the Prevention of Travelers' Diarrhea and Impact on Acquisition of Gut Antimicrobial Resistance Genes
Brief Title: Bismuth Subsalicylate's Role in the Prevention of Travelers' Diarrhea
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to reach target sample size.
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Procter and Gamble (Industry); The New York Center for Travel and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Kristina Angelo, Medical Epidemiologist; Study co-Principal Investigator, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 7082
Record Dates: First submitted 2018-05-01; First posted 2018-05-24 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Diarrhea Travelers; Antibiotic Resistant Infection
MeSH Terms: interventions — bismuth subsalicylate; Dioctyl Sulfosuccinic Acid

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a double-blinded, placebo-controlled randomized clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): Bismuth subsalicylate 4 tablets po bid (2.1 grams total of BSS)
  Interventions: Drug: Bismuth subsalicylate
- Placebo (Placebo Comparator): Placebo oral tablet 4 bid
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Bismuth subsalicylate — We aim to determine if there is a biologic benefit to an intervention (BSS administration) in the acquisition of travelers diarrhea and the acquisition of antimicrobial resistance genes.
  Other Names: Pepto Bismol
  Arms: Intervention Group
Drug: Placebo Oral Tablet — Placebo manufactured to mimic pepto bismol
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the use of prophylactic bismuth subsalicylate (BSS) has an effect on the acquisition of travelers' diarrhea (TD) or antimicrobial resistance (AMR) genes in fecal samples among international travelers who departed from the United States to South East Asia, South Central Asia, or Africa. Our hypotheses will be tested using a double-blinded, placebo controlled randomized clinical trial with participants from a pre-travel health clinic in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 and <70 years of age at the time of enrollment
2. Sign an informed consent stating willingness to participate and comply with the study protocol
3. Plan on leaving for an international trip ≥7 days after their pre-travel consultation
4. Plan on traveling in country for ≥7 days but ≤21 days (21 day limit due to BSS duration recommendations and a lack of data on longer-term BSS use)
5. Traveling to either South East Asia, South Central Asia, North Africa, or Sub-Saharan Africa for at least 7 days of their itinerary
6. Be willing to complete an initial eligibility screening
7. Be willing to complete questionnaires and provide biologic specimens (stool) within 7 days of departure and within 10 days after return
8. Be willing to refrain from taking any pre-biotics, probiotic, synbiotic and/or herbal supplements throughout their study period

Exclusion Criteria:

1. Are <18 years of age or >69 years of age
2. Are traveling in country for <7 or >21 days
3. Have known or suspected contraindications to taking BSS (including, but not limited to, travelers with kidney disease, diabetes, gout, a clotting disorder, or an allergy to any component of BSS)
4. Are pregnant (via self-report), are planning to become pregnant, or may become pregnant during travel (not actively using contraception and are sexually active), or are breastfeeding
5. Routinely take a medication known to interact with BSS (including, but not limited to, insulin, methotrexate, valproic acid, angiotensin-converting enzyme inhibitors, anticoagulants, or other salicylates)
6. Have taken an antibiotic in the 30 days before departure
7. Have taken any medications that may lower one's ability to fight infection (e.g., steroids, monoclonal antibodies, etc.)
8. Have previous diagnoses of immunocompromising conditions such as HIV/AIDS, complement deficiency, immunoglobulin deficiency, or undergoing active chemotherapy or participants with chronic gastrointestinal disorders, such as chronic diarrhea, irritable bowel syndrome (IBS), inflammatory bowel disease (i.e., Crohn's disease, ulcerative colitis), celiac disease, malabsorption syndromes, pancreatic insufficiency, gallbladder disease, or current gastrointestinal cancer
9. Have had diarrhea anytime in the previous 30 days, have diarrhea at the pre-travel consultation, or develop diarrhea before departure
10. Have been given doxycycline for malaria prophylaxis for the current trip (due to possible drug-drug interactions and decreased absorption of the doxycycline)
11. Have an allergy to any component of the placebo tablets

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Connor, MD, Principal Investigator — The New York Center for Travel and Tropical Medicine
Locations (1):
- Marina Rogova, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gibb RD, Brum JM, Sloan KJ, Pitz AM, Circello BT, Grayling RA. Revisiting the efficacy of bismuth subsalicylate for the prevention of traveller's diarrhoea. J Travel Med. 2025 Oct 1;32(6):taaf076. doi: 10.1093/jtm/taaf076. PMID 40720752

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Placebo
Started | 207 | 207
Completed | 136 | 134
Not Completed | 71 | 73
Not completed — Lost to Follow-up | 71 | 73

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Placebo | Total
Number analyzed (Participants) | 136 | 134 | 270
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [27 to 40] | 32 [27 to 45] | 32 [27 to 44]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 51 | 49 | 100
  Female | 84 | 85 | 169
  Missing | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 4 | 16
  Not Hispanic or Latino | 116 | 123 | 239
  Unknown or Not Reported | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 13 | 10 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 32 | 56
  White | 73 | 71 | 144
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 25 | 21 | 46
Region of Enrollment [Number; unit: participants]
  United States | 136 | 134 | 270

OUTCOME MEASURES:

1. Primary Outcome: Traveler's Diarrhea
Description: Self-reported TD
Time Frame: Change from baseline through 10 days post-travel
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Placebo
Number analyzed (Participants) | 136 | 134
Participants | 27 | 26

2. Secondary Outcome: Gut AMR Genes
Description: Pre- and post-travel stools will be tested for the presence/absence of AMR genes
Time Frame: Once within 7 days (before travel); once within 10 days (after travel)
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: From initiation of taking study medication (day 1 of travel to a country of interest) through 7 days after patient travel was completed to country(ies) of interest.
Arm/Group | Intervention Group | Placebo
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/134
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/134
Other Adverse Events (participants affected / at risk) | 0/136 | 0/134

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT03535272/Prot_SAP_001.pdf